CLINICAL TRIAL: NCT06163508
Title: A Long Term Follow-Up Study for Subjects Who Have Received Human Glial Restricted Progenitor Cells (hGRPs; Q-Cells®) (LTFU Study)
Brief Title: A Long Term Follow-Up Study for Subjects Who Have Received Q-Cells
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Greenberg, Benjamin M. Greenberg, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0803
Record Dates: First submitted 2023-11-14; First posted 2023-12-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Transverse Myelitis
MeSH Terms: conditions — Myelitis, Transverse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: 10 microliters of Q cells: 10 microliters of Q cells per site
  Interventions: Drug: Q-Cells®
- Cohort 2: 15 microliters of Q cells: 15 microliters of Q cells per site
  Interventions: Drug: Q-Cells®
- Cohort 3: 20 microliters of Q cells: 20 microliters of Q cells per site
  Interventions: Drug: Q-Cells®

INTERVENTIONS:
Drug: Q-Cells® — Long term observational study of patients who received 1 of 3 different amounts of Q-Cells®.

SUMMARY:
This study is an observational study designed to obtain information on the long-term safety, tolerability, and continued activity of Q-Cells®. The study will follow the participants who previously received Q-Cells® for 10 years.

The goal of this observational study is to learn about the long term effects of Q-Cells® in people with transverse myelitis.

The main objectives the study is to evaluate the safety of patients who have received Q-Cells®.

The secondary goal of the study is to get data about the long-term activity of Q-Cells® over a period of 10 years.

Patients will complete exams, lab tests, imaging, and questionnaires to monitor their safety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been administered Q-Cells® as part of Protocol QTM-101 or other treatment Protocol.
2. Subjects must have the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to collect and use protected health information (PHI) in accordance with national and local subject privacy regulations.

Exclusion Criteria:

1. The study is intended to follow all subjects who have received Q-Cells® without exception.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must have been administered Q-Cells® as part of Protocol QTM-101 or other treatment Protocol.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | through study completion, an average of 10 years
  Safety will be assessed by the number of Adverse events.These will be recorded via physical examination findings and will be presented in data listings.
  Clinically significant changes on physical exam in the areas of: general appearance, head, ears, eyes, nose, throat, neck, chest and lungs, cardiovascular, abdomen, neurological, thyroid, musculoskeletal, lymph nodes, extremities and skin, and operative site will be recorded as Adverse Events.
Safety: Vital signs: Systolic Blood Pressure | through study completion, an average of 10 years
  Systolic Blood Pressure: Criteria for Clinically Relevant Vital Signs Abnormalities: >180 mmHg or an increase from pre-dosing of more than 40 mmHg, or <90 mmHg or a decrease from pre-dosing of more than 30 mmHg
Safety Endpoints: Vital signs: Diastolic Blood Pressure | through study completion, an average of 10 years
  Diastolic Blood Pressure: Criteria for Clinically Relevant Vital Signs Abnormalities: >105 mmHg or an increase from pre-dosing of more than 30 mmHg, or <50 mmHg or a decrease from pre-dosing of more than 20 mmHg
Safety Endpoints: Vital signs: Pulse | through study completion, an average of 10 years
  Pulse: Criteria for Clinically Relevant Vital Signs Abnormalities: >120 beats per minute or an increase from pre dosing of more than 20 beats per minute, or <50 beats per minute or a decrease from pre dosing of more than 20 beats per minute
Safety Endpoints: Vital signs: Temperature | through study completion, an average of 10 years
  Temperature: Criteria for Clinically Relevant Vital Signs Abnormalities: >38.5°C and an increase from pre-dosing of at least 1°C
Safety as measured by change in Electrocardiogram (ECG) measures from baseline at 10 years | through study completion, an average of 10 years (Baseline, 10 years)
  Number of participants with abnormal ECG readings will be summarized using descriptive statistics by original treatment cohort and visit. ECG findings that are determined to be potentially clinically significant will be summarized.
Safety Endpoints: Clinical Laboratory assessments: chemistry | through study completion, an average of 10 years
  Descriptive statistics for raw values as well as change from baseline (entry into this protocol No. QLTFU-101) by original treatment group will be presented for each visit. The number and percentage of subjects with potentially clinically significant laboratory results will be tabulated by original treatment cohort and overall.
Safety Endpoints: Clinical Laboratory assessments: hematology | through study completion, an average of 10 years
  Descriptive statistics for raw values as well as change from baseline (entry into this protocol No. QLTFU-101) by original treatment group will be presented for each visit. The number and percentage of subjects with potentially clinically significant laboratory results will be tabulated by original treatment cohort and overall.

SECONDARY OUTCOMES:
Exploratory Endpoints: Visual Analog pain Scale (VAS) | through study completion, an average of 10 years
  Changes in pain will be assessed using VAS, a self-assessment where patients rank their current pain from 0-10.
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: American Spinal Injury Association (ASIA) Impairment Scale | through study completion, an average of 10 years
  Neurological changes in muscle strength and sensation via the ASIA exam.
  ASIA exam yields overall scores ranked alphabetically A through E where A is the most impaired and E is normal.
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life Questionnaire: Lower Extremity Function (mobility) | through study completion, an average of 10 years
  NIH PROMIS scale for Lower Extremity Function is a self-assessment where patients score their lower extremity function. Higher scores in this scale are related to better outcomes.
  Minimum value: 95 Maximum value: 19
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life Questionnaire: Neurogenic Bladder Symptom Score (NBSS) | through study completion, an average of 10 years
  NIH PROMIS scale for NBSS is a self-assessment where patients score their bladder symptoms. Lower scores in this scale are related to better outcomes.
  Minimum value: 28 Maximum value: 0
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life Questionnaire: Neurogenic Bowel Dysfunction | through study completion, an average of 10 years
  NIH PROMIS scale for Neurogenic Bowel Dysfunction is a self-assessment where patients score their bowel symptoms. Lower scores in this scale are related to better outcomes.
  Minimum value: 47 Maximum value: 0
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life Questionnaire: Erectile Function | through study completion, an average of 10 years
  NIH PROMIS scale for Erectile Function is a self-assessment where patients score their sexual function. Higher scores in this scale are related to better outcomes.
  Minimum value: 5 Maximum value: 53
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.
Neurological change: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Quality of Life Questionnaire: Sexual Function | through study completion, an average of 10 years
  NIH PROMIS scale for Sexual Function is a self-assessment where patients score their sexual function. Lower scores in this scale are related to better outcomes.
  Minimum value: 0 Maximum value: 263
  Analysis of activities is considered exploratory and observational data from each patient will be recorded due to sample size.
  Descriptive statistics (N, mean, standard deviation, median, minimum and maximum values) and change from baseline will be summarized overall and by original treatment cohort and visit.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, MD, Principal Investigator — University of Texas Southwestern Medial Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided